A Cohort Study of Weight Loss and Gliosis NCT0357887 6/9/2025

## Statistical Analysis Plan

Weight loss will be determined by the percentage change in weight during the 6-month behavioral weight loss program. For all participants, weight change will be calculated as weight at 6-months minus weight at baseline, as a percentage. Weight regain will be considered during the 12-month follow up period. Change in kilograms of weight will be calculated from the 18-month visit minus weight at the 6-month visit. Weight change outcomes will be tested by One-way ANOVA with Bonferroni correction for multiple comparisons. P-values less than 0.05 will be considered significant. Analyses will be unadjusted.